CLINICAL TRIAL: NCT06469255
Title: Effects of Short-Term Low-Calorie Ketogenic Diet on Biochemical and Anthropometric Parameters in Women With Polycystic Ovary Syndrome
Brief Title: Short Term Ketogenic Diet in Polycictic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hande Seven Avuk, Head of Nutrition and Dietetic Department, Clinical Assistant Professor, Istanbul Bilgi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDPCOS; 2019-14/17 (Registry Identifier: Acıbadem Mehmet Ali Aydınlar University on Medical Research Evaluation Board)
Record Dates: First submitted 2024-03-12; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Obesity; Menstrual Dysfunction; Ketogenic Diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet Intervention (Experimental): 4 weeks low calorie Ketogenic Diet intervention
  Interventions: Other: Diet Treatment

INTERVENTIONS:
Other: Diet Treatment — 4 weeks low calorie diet treatment

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common health problems in women of reproductive age, characterized by increased androgen levels, impaired ovulatory functions, and polycystic ovaries. In addition to cosmetic problems including hirsutism and acne, it also poses a risk for significant chronic diseases, including infertility, dyslipidemia, obesity, sleep apnea, diabetes, cardiovascular diseases, and various malignancies.

The aim of this clinical study was to investigate the effects of short-term low-calorie ketogenic diet (LCKD) intervention on anthropometric, biochemical and hormonal parameters in women with PCOS. The main questions it aims to answer are:

* Is a short-term low-calorie ketogenic diet effective on body composition in overweight women with PCOS?
* Is a short-term low-calorie ketogenic diet effective on biochemical and hormonal parameters in overweight women with PCOS?

Participants were diagnosed with PCOS according to the Rotterdam 2003 criteria as a result of the clinical, biochemical and ultrasonographic medical evaluation made by the gynecologist, and those who were found to be eligible for LCKD and volunteered to participate in the study were included in the study.

Researchers are examining whether a low-calorie ketogenic diet applied between two menstrual cycles has any effects on anthropometric, biochemical and hormonal parameters in women with PCOS.

DETAILED DESCRIPTION:
This study was conducted on patients who applied to a nutrition and diet consultancy center in İstanbul.All patients provided written informed consent before the start of the study and after receiving a detailed explanation of the procedures. The sample size of this study was that of Paoli et al. (19) according to the reference study were taken as d: 1.737 and SD: 2.1 for the change parameter observed in the BMI level, and with a 95% confidence interval,1-β: 0.95 and α: 0.05 were determined as at least 7 individuals in the G*Power program.

Exclusion Criteria: Those with any endocrine disorders other than PCOS, chronic liver or kidney disease, hypertension, hyperuricemia, heart failure, infarction or cerebrovascular disease, pregnant and breastfeeding women, those with severe psychiatric disorders, oncological diseases, those using medications that may affect biochemical parameters, and individuals with special dietary needs were excluded in this study.

General Plan of the Study: During the study, four follow-up interviews were held at 7-10-day intervals to monitor participants' diet compliance and body composition changes.During the first meeting, information was provided verbally and in writing regarding the purpose and scope of the study, and an informed consent form was signed. The second interview was held on the second or third day of menstruation. During this meeting, blood was taken from the individuals to analyze biochemical parameters, and then their anthropometric measurements were taken and LCKD was given. Additionally, to determine whether LCKD was not applied before the intervention, a urine ketone test was performed, wherein urine samples were examined for the presence of ketones. During the third interview, urine ketone test was performed to evaluate participants' compliance with the diet, and body composition changes were monitored. During the study, to track their food consumption, participants shared photos of the meals they consumed with the researcher. The fourth and final interview was conducted on the second or third day of the first menstrual period after the LCKD intervention started. The presence of ketosis was determined by examining the urine ketone level again. Subsequently, blood was taken for basal hormone and biochemical measurements, anthropometric measurements were evaluated for the last time, and the LCKD intervention was completed.This intervention study was conducted between two menstrual cycles.

Planning a Ketogenic Diet Intervention: A personalized LCKD was planned. Daily energy requirement is the sum of basal metabolic rate, physical activity factor (1.4), and thermal energy of food (10%). Mifflin-St. Joer's equation was used to determine the basal metabolic rate. Total daily energy requirement was reduced by 500 calories. Castellana et al. suggested that the macronutrient content of the LCKD was calculated as carbohydrates of <20 g/day and protein of 0.8-1.2 g/kg/day. It is calculated according to the individuals' carbohydrate and protein needs, with the remainder of the total energy coming from fat. Daily fat consumption is >30-40 g/day, as in typical LCKDs (Castellana et al., 2020). Participants were allowed to eat unlimited green leafy vegetables, cruciferous vegetables, squash, and cucumbers during the intervention.

This study was conducted on patients who applied to a nutrition and diet consultancy center in İstanbul.All patients provided written informed consent before the start of the study and after receiving a detailed explanation of the procedures. The sample size of this study was that of Paoli et al. (19) according to the reference study were taken as d: 1.737 and SD: 2.1 for the change parameter observed in the BMI level, and with a 95% confidence interval,1-β: 0.95 and α: 0.05 were determined as at least 7 individuals in the G*Power program.

Exclusion Criteria: Those with any endocrine disorders other than PCOS, chronic liver or kidney disease, hypertension, hyperuricemia, heart failure, infarction or cerebrovascular disease, pregnant and breastfeeding women, those with severe psychiatric disorders, oncological diseases, those using medications that may affect biochemical parameters, and individuals with special dietary needs were excluded in this study.

General Plan of the Study: During the study, four follow-up interviews were held at 7-10-day intervals to monitor participants' diet compliance and body composition changes.During the first meeting, information was provided verbally and in writing regarding the purpose and scope of the study, and an informed consent form was signed. The second interview was held on the second or third day of menstruation. During this meeting, blood was taken from the individuals to analyze biochemical parameters, and then their anthropometric measurements were taken and LCKD was given. Additionally, to determine whether LCKD was not applied before the intervention, a urine ketone test was performed, wherein urine samples were examined for the presence of ketones. During the third interview, urine ketone test was performed to evaluate participants' compliance with the diet, and body composition changes were monitored. During the study, to track their food consumption, participants shared photos of the meals they consumed with the researcher. The fourth and final interview was conducted on the second or third day of the first menstrual period after the LCKD intervention started. The presence of ketosis was determined by examining the urine ketone level again. Subsequently, blood was taken for basal hormone and biochemical measurements, anthropometric measurements were evaluated for the last time, and the LCKD intervention was completed.This intervention study was conducted between two menstrual cycles.

Planning a Ketogenic Diet Intervention: A personalized LCKD was planned. Daily energy requirement is the sum of basal metabolic rate, physical activity factor (1.4), and thermal energy of food (10%). Mifflin-St. Joer's equation was used to determine the basal metabolic rate. Total daily energy requirement was reduced by 500 calories. Castellana et al. suggested that the macronutrient content of the LCKD was calculated as carbohydrates of <20 g/day and protein of 0.8-1.2 g/kg/day. It is calculated according to the individuals' carbohydrate and protein needs, with the remainder of the total energy coming from fat. Daily fat consumption is >30-40 g/day, as in typical LCKDs (Castellana et al., 2020). Participants were allowed to eat unlimited green leafy vegetables, cruciferous vegetables, squash, and cucumbers during the intervention.

Food Consumption Evaluation: Participants' food consumption before the dietary intervention was recorded using the 24-h reminder method (2 days on weekdays and 1 day on the weekend).

Biochemical Measurements:This study was conducted between two menstrual cycles to accurately determine baseline and ending basal hormone levels, and biochemical parameters were measured by blood collection on the second to third day of menstruation. On the following days, a nurse extracted blood samples following an 8-12-h fasting. Subsequently, the blood samples were examined for fasting insulin, fasting blood glucose, total cholesterol, triglyceride, HDL-cholesterol, LDL-cholesterol, DHEA-SO4, androstenedione, LH, FSH, estradiol, SHBG, total testosterone, prolactin, IGF-1, and TNF-α levels. HOMA-IR, which was developed by Mathews et al., was used to determine insulin resistance using fasting glucose and insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals who were diagnosed with PCOS according to the Rotterdam 2003 criteria,
* Individuals suitable for LCKD

Exclusion Criteria:

* Endocrine disorders other than PCOS,
* Chronic liver disease,
* Chronic kidney disease,
* Hypertension,
* Hyperuricemia,
* Heart failure, infarction or cerebrovascular disease,
* Pregnant and breastfeeding women,
* Severe psychiatric disorders,
* Oncological diseases,
* Individuals using medications that may affect biochemical parameters,
* Individuals with special dietary needs

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Polycystic ovary syndrome patients
Enrollment: 13 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Anthropometric Measurements - Body weight and composition | 4 weeks (Between two menstrual cycle)
  Body weight (kg) of the participants were measured in light clothing on an empty stomach, following anthropometric measurement standards (Norton, 2018). Total body weight and body composition analysis (fat ratio, fat, muscle, fluid mass, and phase angle [PhA]) were performed following the protocol using the TANİTA MC780 MA bio-electrical impedance device with a sensitivity of 50 grams.
Anthropometric Measurements - Height | 4 weeks (Between two menstrual cycle)
  Height (cm) measurements of the participants were measured following anthropometric measurement standards with stadiometer (Norton, 2018).
Anthropometric Measurements - Circumferences | 4 weeks (Between two menstrual cycle)
  Waist, hip, neck, upper middle arm, and chest circumference measurements of the participants were measured in light clothing on an empty stomach, following anthropometric measurement standards (Norton, 2018).
Body Mass Index | 4 weeks (Between two menstrual cycle)
  Body mass index (BMI) (kg/m2) was calculated using the following equation: body weight (kg)/height (m2) (Misra & Dhurandhar, 2019).
Biochemical Measurements | 4 weeks (Between two menstrual cycle)
  This study was conducted between two menstrual cycles to accurately determine baseline and ending basal hormone levels, and biochemical parameters were measured by blood collection on the second to third day of menstruation. On the following days, a nurse extracted blood samples following an 8-12-h fasting. Subsequently, the blood samples were examined for fasting insulin, fasting blood glucose, total cholesterol, triglyceride, HDL-cholesterol, LDL-cholesterol, DHEA-SO4, androstenedione, LH, FSH, estradiol, SHBG, total testosterone, prolactin, IGF-1, and TNF-α levels. HOMA-IR, which was developed by Mathews et al., was used to determine insulin resistance using fasting glucose and insulin levels. It is calculated using the following formula: HOMA-IR = (fasting glucose [mg/dL] × fasting insulin [uIU/mL])/405 (Matthews et al., 1985).

SECONDARY OUTCOMES:
Food Consumption Evaluation | 1 times before intervention
  Participants' food consumption before the dietary intervention was recorded using the 24-h reminder method (2 days on weekdays and 1 day on the weekend). Intakes of macro- and micronutrients such as energy, carbohydrates, proteins, and fats were evaluated using the Nutrition Information System (BeBİS) 8.2 full version program (BeBİS, 2019).

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paoli A, Mancin L, Giacona MC, Bianco A, Caprio M. Effects of a ketogenic diet in overweight women with polycystic ovary syndrome. J Transl Med. 2020 Feb 27;18(1):104. doi: 10.1186/s12967-020-02277-0. PMID 32103756
- [Background] Mavropoulos JC, Yancy WS, Hepburn J, Westman EC. The effects of a low-carbohydrate, ketogenic diet on the polycystic ovary syndrome: a pilot study. Nutr Metab (Lond). 2005 Dec 16;2:35. doi: 10.1186/1743-7075-2-35. PMID 16359551
- [Background] Barber TM, Franks S. Obesity and polycystic ovary syndrome. Clin Endocrinol (Oxf). 2021 Oct;95(4):531-541. doi: 10.1111/cen.14421. Epub 2021 Jan 31. PMID 33460482
- [Background] Barrea L, Verde L, Camajani E, Cernea S, Frias-Toral E, Lamabadusuriya D, Ceriani F, Savastano S, Colao A, Muscogiuri G. Ketogenic Diet as Medical Prescription in Women with Polycystic Ovary Syndrome (PCOS). Curr Nutr Rep. 2023 Mar;12(1):56-64. doi: 10.1007/s13668-023-00456-1. Epub 2023 Jan 25. PMID 36695999
- [Background] Cincione RI, Losavio F, Ciolli F, Valenzano A, Cibelli G, Messina G, Polito R. Effects of Mixed of a Ketogenic Diet in Overweight and Obese Women with Polycystic Ovary Syndrome. Int J Environ Res Public Health. 2021 Nov 27;18(23):12490. doi: 10.3390/ijerph182312490. PMID 34886216
- [Background] Fauser BC, Tarlatzis BC, Rebar RW, Legro RS, Balen AH, Lobo R, Carmina E, Chang J, Yildiz BO, Laven JS, Boivin J, Petraglia F, Wijeyeratne CN, Norman RJ, Dunaif A, Franks S, Wild RA, Dumesic D, Barnhart K. Consensus on women's health aspects of polycystic ovary syndrome (PCOS): the Amsterdam ESHRE/ASRM-Sponsored 3rd PCOS Consensus Workshop Group. Fertil Steril. 2012 Jan;97(1):28-38.e25. doi: 10.1016/j.fertnstert.2011.09.024. Epub 2011 Dec 6. PMID 22153789
- [Background] Misra A, Dhurandhar NV. Current formula for calculating body mass index is applicable to Asian populations. Nutr Diabetes. 2019 Jan 28;9(1):3. doi: 10.1038/s41387-018-0070-9. No abstract available. PMID 30692514
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- See also: Norton, K. I. (2018). Standards for anthropometry assessment. In Kinanthropometry and exercise physiology (pp. 68-137). Routledge. — https://www.researchgate.net/publication/333585249_Standards_for_Anthropometry_Assessment